CLINICAL TRIAL: NCT03485144
Title: A Phase II Randomized, Double-blinded, Placebo-controlled Clinical Study to Evaluate the Immunogenicity and Safety of TetraVax-DV in Healthy Adults in Taiwan
Brief Title: A Clinical Study to Evaluate TV003 in Healthy Adults in Taiwan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT-DV-21
Record Dates: First submitted 2018-03-02; First posted 2018-04-02 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TV003 (Experimental): Live Attenuated Virus Vaccine-TetraVax-DV
  Interventions: Biological: TV003
- Placebo for TV003 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo for TV003

INTERVENTIONS:
Biological: TV003 — Live attenuated virus vaccine-TetraVax-DV
  Arms: TV003
Biological: Placebo for TV003 — Placebo
  Arms: Placebo for TV003

SUMMARY:
The goal of this study is to determine the immunogenicity and safety of TV003(TetraVax-DV), a live attenuated tetravalent dengue vaccine candidate, in healthy human subjects in Taiwan

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 20 and 70 years of age
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study
* Willingness to sign the informed consent document
* Female of childbearing potential willing to use effective contraception for the duration of the trial

Exclusion Criteria:

* Females currently pregnant, as determined by positive β- human choriogonadotropin (HCG) test, and/or breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease
* Below lower limit of normal for absolute neutrophil count
* Any significant alcohol or drug abuse in the past 12 months
* History of a severe allergic reaction or anaphylaxis
* Self-reported systemic hypersensitivity to any of the vaccine components
* Severe asthma
* Known HIV, Hepatitis B or hepatitis C
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Receive chronic administration of immunosuppressant drugs within 6 months prior to the administration of the study vaccine
* Use of any investigational product within 30 days before study vaccination or at any time during the study
* Asplenia
* Receive administration of immunoglobulins and/or any blood products within 12 months preceding the administration of the study vaccine or at any time during the study
* Fever or suspected fever within 72 hours prior to vaccination or tympanic temperature greater than 38°C on the day of vaccination
* Receive administration of any licensed live attenuated vaccines within 30 days preceding the administration of the study vaccine and ending 30 days after
* Receive administration of any licensed inactivated vaccines within 14 days preceding the administration of the study vaccine and ending 14 days after
* Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of TetraVax-DV assessed by plaque reduction neutralization titer 50% (PRNT50) | Up to Day 90 after vaccination
  Determination of the serum PRNT50 to each virus type for each subject at study day 28, 56 and 90 post vaccination.

SECONDARY OUTCOMES:
Immunogenicity of TetraVax-DV assessed by response rates | Up to Day 90 after vaccination
  Determine monovalent, bivalent, trivalent, and tetravalent seropositivity and seroconversion rates.
Duration of immunogenicity of TetraVax-DV assessed by PRNT50 | Up to Day 365 after vaccination
  Assess the duration of the antibody response by measured serum PRNT50 to each virus type for each subject at study day 180 and day 365 post vaccination.
Frequency of viremia following vaccination | Up to Day 15 after vaccination
Quantity of viremia following vaccination | Up to Day 15 after vaccination
Duration of viremia following vaccination | Up to Day 15 after vaccination
Determine the number of vaccinees with recoverable dengue virus. | Up to Day 15 after vaccination
Determine the safety of TetraVax-DV assessed by frequency of solicited local adverse reactions. | Up to Day 7 after vaccination.
Determine the safety of TetraVax-DV assessed by frequency of solicited systemic and unsolicited adverse reactions. | Up to Day 21 after vaccination.
Determine the safety of TetraVax-DV assessed by occurrence of adverse events and serious adverse events. | Up to Day 365 after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan